CLINICAL TRIAL: NCT03427476
Title: CTT1057, a Small Molecular Inhibitor of Prostate Specific Membrane Antigen (PSMA), as a Novel Imaging Agent of Neovascularization in Renal Cell Carcinoma (RCC): A Pilot Study
Brief Title: CTT1057, a Small Molecular Inhibitor of PSMA, as a Novel Imaging Agent of Neovascularization in Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Targeted Technology (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1057-102
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-01

CONDITIONS: Renal Cell Carcinoma
Keywords: renal cell carcinoma; RCC; prostate specific membrane antigen; PSMA; metastatic renal cancer; positron emission tomography; PET
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metastatic RCC (> 3 lesions) (Experimental): Patients with metastatic renal cell carcinoma and planned biopsy of a metastatic lesion (N = 5)
  Interventions: Drug: CTT1057
- RCC patients with primary lesions > 7 mm in diameter (Experimental): Cohort B: Patients with evidence of primary renal cell carcinoma and lesions > 7 cm (may also have metastatic disease) (N = 5)
  Interventions: Drug: CTT1057

INTERVENTIONS:
Drug: CTT1057 — Cohort A: Single IV dose (370 MBq, or 10 mCi). Combined PET/MR or PET/CT imaging (kidney + whole body) will be performed following tracer injection. Patients in cohort A will undergo metastatic lesion biopsy (plus lymph node dissection) within 12 weeks after CTT1057 PET.
  Cohort B: Single IV dose (370 MBq, or 10 mCi). Combined PET/MR or PET/CT imaging (kidney + whole body) will be performed following tracer injection. Patients in cohort B (renal cell carcinoma) will have nephrectomy within 12 weeks of CTT1057 PET imaging.

SUMMARY:
The purpose of this study is to test a novel diagnostic PET imaging agent for safety and biodistribution. The agent binds PSMA and is designed to detect Prostate Specific Membrane Antigen expressing tumors, such as has been described for some renal cell carcinoma tumors.

DETAILED DESCRIPTION:
CTT has developed a PET imaging agent, CTT1057, labeled with 18F, that is based on a small molecule core and targets an extracellular region of PSMA with high affinity. Although comparable to other inhibitors in terms of affinity for PSMA, this unique class of phosphoramidate agents are the only known irreversible PSMA inhibitors. Due to its irreversible binding to PSMA and rapid uptake by PSMA-expressing cancer cells, accumulation at the cancer target is expected to be rapid, specific and sensitive. PSMA expression has been reported in renal cell carcinoma cells, making it possible that CTT1057 may have utility in detecting these tumors.

Ten patients will be enrolled in parallel in two cohorts:

* (Cohort A) Patients with presumed metastases on conventional imaging, with at least one presumed metastatic lesion measuring > 1.5 cm in diameter (long-axis for non-node target lesions; short axis for lymph node), with planned biopsy of a metastatic lesion (N = 5).
* (Cohort B) Patients with primary renal mass measuring > 7 cm on conventional imaging, with presumptive or histologically confirmed diagnosis of renal cell carcinoma, with planned nephrectomy. Patients may or may not have nodal or distant metastases on conventional imaging (N = 5) Participants receive a single IV dose (370 MBq, or 10 mCi) of CTT1057 in this trial. Combined PET/MR or PET/CT imaging (kidney + whole body) will be performed following tracer injection. Patients in cohort A (metastatic renal cell carcinoma) will undergo planned metastatic lesion biopsy within 12 weeks following CTT1057 PET imaging. Patients in cohort B (primary renal cell carcinoma) will have planned nephrectomy within 12 weeks following CTT1057 PET imaging.

The one-time nominal injected dose will be 370 MBq (10 mCi). Estimated mass dose is 20 µg of CTT1057. Dose will be in a volume of 3 - 5 mL, and will be injected intravenously as a bolus injection.

Vital signs, adverse event assessment, and 12 lead ECGs will be performed on day 1 before and after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years old
* Histologically confirmed renal cell carcinoma
* Adequate organ function including:
* - Platelet count of > 50,000/mm3
* - Neutrophil count of > 1000/mm3
* - Serum Cr < 1.5 x ULN or estimated GFR > 60 ml/min based upon Cockroft-Gault equation
* - Proteinuria < 1 g/24 hours based upon 24 hour urine collection or spot urine protein/creatinine ratio
* - AST and ALT < 2.5 x ULN (< 5 x ULN in patients with known liver metastases)
* - Total bilirubin < 1.5 x ULN (< 3 x ULN in patients with known/suspected Gilbert's disease)
* ECOG performance status of 0 or 1
* Able to provide written informed consent and willing to comply with protocol requirements
* No contra-indication to MR including severe claustrophobia, incompatible aneurysm clips or cardiac pacemaker
* For participants of childbearing potential, not pregnant, and use of effective contraceptive methods during the trial and within 6 months following radiotracer injection
* Cohort A only: Presence of at least three distinct metastatic lesions by standard imaging including whole body bone scan + cross-sectional imaging of the abdomen and pelvis obtained within 12 weeks prior to protocol scan
* Cohort B only: (N = 5 evaluable patients): Planned nephrectomy within 12 weeks following protocol scan

Exclusion Criteria:

* Patients with or with a history of uncontrolled bleeding diathesis
* Inadequate venous access per assessment of treating health care provider
* Receipt of radioisotope within 5 physical half-lives prior to trial enrollment
* Prior treatment with alpha radiation therapy (Radium Ra 223 chloride; Xofigo™) during the previous 60 days
* Have a medical condition or other circumstances that, in the opinion of the investigator would significantly decrease the chances of obtaining reliable data, achieving the study objectives, or completing the trial.
* Prior history of any other malignancy within past three years, except melanomatous skin cancer or carcinoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse event frequency as graded by Common Toxicity Criteria version 4.03 | 7 days from time of injection

SECONDARY OUTCOMES:
CTT1057 detection in blood samples | Up to four hours from time of injection
Compare the level of CTT1057 uptake on PET imaging of localized renal cell carcinoma with PSMA protein expression by immunohistochemistry from subsequent nephrectomy specimens | 12 weeks
Standardized Uptake Value (SUV) of CTT1057 PET for positive and negative tumor pathology results from primary renal cell carcinoma lesion tissue | 4 hours
Lesion-by-lesion basis tracer sensitivity ans specificity compared with standard imaging in metastatic renal cell carcinoma | 4 hours
Identification of positive lesions on CTT1057 PET in subjects with equivocal or negative conventional imaging scans | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Langton-Webster, PhD, Study Chair — Cancer Targeted Technology
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided